CLINICAL TRIAL: NCT03789110
Title: NIMBUS: A Phase II Study of Nivolumab Plus Ipilimumab in Metastatic Hypermutated HER2-negative Breast Cancer
Brief Title: NIMBUS: Nivolumab Plus Ipilimumab in Metastatic Hypermutated HER2-negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Sara Tolaney, MD, Primary Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-561
Record Dates: First submitted 2018-12-26; First posted 2018-12-28 (Actual); Results first posted 2022-09-27 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab+Ipilimumab (Experimental): * Ipilimumab is administered intravenously every 6 weeks
  * Nivolumab is administered intravenously every 2 weeks
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is called an anti- PD-1 or a checkpoint inhibitor and is an antibody (a type of human protein) designed to allow the body's own immune system to destroy tumors
  Other Names: Opdivo
Drug: Ipilimumab — Ipilimumab is called an anti-CTLA-4 and is a type of antibody that works to prevent the body's immune system from stopping to fight a specific cancer
  Other Names: Yervoy

SUMMARY:
This research study is studying a drug combination of nivolumab and ipilimumab as a possible treatment for hypermutated HER2 negative breast cancer.

The drugs involved in this study are:

* Nivolumab (Opdivo ®)
* Ipilimumab (Yervoy ®)

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

Nivolumab is called an anti- PD-1 or a checkpoint inhibitor and is an antibody (a type of human protein) designed to allow the body's own immune system to destroy tumors. Ipilimumab is called an anti-CTLA-4 and is a type of antibody that works to prevent your body's immune system from stopping to fight this specific cancer.

The U.S. Food and Drug Administration (FDA) has not approved nivolumab for this specific disease but it has been approved for other uses including but not limited to non-small cell lung cancer, melanoma and renal cell carcinoma.

The U.S. Food and Drug Administration (FDA) has not approved ipilimumab for this specific disease but it has been approved for other uses such as melanoma and renal cell carcinoma.

The combination of nivolumab with ipilimumab may or may not increase anti-cancer activity by further boosting the immune system. At this time, the FDA has not approved nivolumab in combination with ipilimumab for this specific disease although these drugs have been approved for other uses such as melanoma and renal cell carcinoma.

The purpose of this research study is to determine how nivolumab together with ipilimumab, works in treating breast cancer that has spread to other parts of the body. The investigators are also investigating whether there are certain DNA or protein markers in the blood or tumor tissue that may indicate whether the combination will work in future patients

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed invasive breast cancer, with metastatic disease. Participants without pathologic or cytologic confirmation of metastatic disease should have unequivocal evidence of metastasis from physical examination or radiologic evaluation.
* Breast cancer must be HER2-negative by IHC or non-amplified as determined by the current ASCO-CAP criteria. If patient has more than one histological result, the most recent one will be usedfor inclusion. Participants may be ER/PR positive or negative.
* Patients must harbor tumors with total mutational burden (TMB) of at least 9 mutations per megabase assessed by a cancer-gene panel containing more than 300 genes, and performed in a CLIA verified laboratory. Tests like Foundation One, Oncopanel (DFCI), or IMPACT (MSKCC) are acceptable for including patients on this trial.
* Participants must have measurable disease by RECIST version 1.1.
* Participants must agree to undergo a research biopsy, if tumor is safely accessible, at baseline and at day 29 cycle 1 (+14 scheduling window). Previously collected archival tissue will be obtained on all participants. Participants for whom newly-obtained samples cannot be provided (e.g. inaccessible or participant safety concern) may submit an archived specimen (block or if not possible, 20 unstained slides).
* Prior chemotherapy: Participants may have received 0-3 prior chemotherapeutic regimens for metastatic breast cancer and must have been off treatment with chemotherapy for at least 14 days prior to study treatment initiation.
* Patients with hormone receptor positive breast cancer must have progressed on at least one prior line of endocrine therapy in the metastatic setting or have disease recurrence while on adjuvant endocrine therapy.
* Participants should also be adequately recovered from acute toxicities of prior treatment, with the exception of alopecia and peripheral sensory neuropathy.
* Prior biologic therapy: Patients must have discontinued all biologic therapy at least 14 days prior to study treatment initiation.
* Prior radiation therapy: Patients may have received prior radiation therapy in either the metastatic or early-stage setting. Radiation therapy must be completed 14 days prior to study treatment initiation.
* In all cases, there must be no ongoing complications from prior radiotherapy.
* The subject is ≥18 years old.
* ECOG performance status ≤1(Karnofsky ≥70%, see Appendix A).
* Participants must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,000/mcL
  * platelets ≥100,000/mcL
  * hemoglobin ≥ 8 g/dl
  * total bilirubin ≤1.5 × institutional upper limit of normal (ULN) (or ≤ 2.0 x ULN in patients with documented Gilbert's Syndrome)
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN or (≤ 3 × institutional ULN for participants with documented liver metastases)
  * creatinine ≤1.5 × institutional ULN OR creatinine clearance ≥ 40 mL/min (using Cockcroft-Gault formula) for participants with creatinine levels above institutional ULN.
* Female subjects of childbearing potential must have a negative pregnancy test (serum or urine) at screening.
* Childbearing potential is defined as: participants who have not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause) and has not undergone surgical sterilization (removal of ovaries and/or uterus).
* Female and male participants of childbearing potential must agree to use an adequate method of contraception. For women, contraception is required starting with the first dose of study medication through 150 days (5 months) after the last dose of study medication. For men who are sexuall active with women of childbearing potential, contraception is required starting with the first dose of study medication for a period of 7 months after the last dose of nivolumab. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established and proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* Participants on bisphosphonates may continue receiving bisphosphonate therapy during study treatment. Initiation of bisphosphonate or RANKL agent is allowed on study.
* The participant is capable of understanding and complying with the protocol and has signed the informed consent document.

Exclusion Criteria:

* Major surgery within 2 weeks before the first dose of study treatment.
* Concurrent administration of other anti-cancer therapy within 14 days of starting protocol therapy and during the course of this study.
* The participant has received another investigational agent within 14 days of the first dose of study drug.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody.
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms. Participants with a history of treated central nervous system (CNS) metastases are eligible. Treated brain metastases are defined as those having no evidence of progression for ≥ 2 weeks after treatment, and no ongoing requirement for corticosteroids, as ascertained by clinical examination and brain imaging (magnetic resonance imaging or CT scan) completed during screening. Subject must be either off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily (or equivalent) for at least 7 days prior to first study treatment. Treatment for brain metastases may include whole brain radiotherapy, radiosurgery, or a combination as deemed appropriate by the treating physician. Participants with CNS metastases treated by neurosurgical resection or brain biopsy performed within 28 days before study treatment initiation will be excluded.
* The subject has uncontrolled, significant intercurrent or recent illness. Individuals with a history of different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years or are deemed by the investigator to be at low risk for recurrence of that malignancy.
* Participant has an active infection requiring IV antibiotics at initiation of study therapy.
* Patient has a medical condition that requires chronic systemic steroid therapy or on any other form of immunosuppressive medication. For example, participants with autoimmune disease that requires systemic steroids or immunosuppression agents should be excluded. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Subjects with current pneumonitis, or requiring supplementary O2 therapy.
* The participant is known to be positive for human immunodeficiency virus (HIV), HepBsAg, or HCV RNA. HIV-positive participants on combination antiretroviral therapy are ineligible
* Participants with any other active malignancy requiring concurrent intervention.
* Known hypersensitivity to any of the components of ipilimumab or nivolumab.
* The participant has received a live vaccine within 28 days prior to the first dose of trial treatment and while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine. The use of the inactivated seasonal influenza vaccine (Fluzone®) is allowed.
* The participant is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2026-02-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tolaney, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Requests may be directed to: [contact information for Sponsor- Investigator or designee]

REFERENCES:
- [Derived] Barroso-Sousa R, Zanudo JGT, Li T, Reddy SM, Emens LA, Kuntz TM, Silva CAC, AlDubayan SH, Chu H, Overmoyer B, Lange P, DiLullo MK, Montesion M, Kasparian J, Hughes ME, Attaya V, Basta A, Lin NU, Tayob N, Jeselsohn R, Mittendorf EA, Tolaney SM. Nivolumab plus low-dose ipilimumab in hypermutated HER2-negative metastatic breast cancer: a phase II trial (NIMBUS). Nat Commun. 2025 May 13;16(1):4430. doi: 10.1038/s41467-025-59695-1. PMID 40360544

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab+Ipilimumab: * Ipilimumab is administered intravenously every 6 weeks
  * Nivolumab is administered intravenously every 2 weeks
  Nivolumab: Nivolumab is called an anti- PD-1 or a checkpoint inhibitor and is an antibody (a type of human protein) designed to allow the body's own immune system to destroy tumors
  Ipilimumab: Ipilimumab is called an anti-CTLA-4 and is a type of antibody that works to prevent the body's immune system from stopping to fight a specific cancer
Period: Overall Study
Arm/Group | Nivolumab+Ipilimumab
Started | 30
Completed | 0
Not Completed | 30
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2
Not completed — Lack of Efficacy | 22
Not completed — still on treatment | 3

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 63 [36 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
ECOG Performance Status [Count of Participants; unit: Participants] — The ECOG (Eastern Cooperative Oncology Group) Scale of Performance Status describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). This is a numbering scale of 0 to 5. The higher the number, the worse the performance status. Zero (0) refers to being full active. 5 is dead.
  Participants
    0 | 22
    1 | 8
Hormone Receptor (HR) Status [Count of Participants; unit: Participants] — HR+ is defined as ER (Estrogen receptors) positive, or PR (progesterone receptors) positive, or Her2 positive Triple negative is defined as ER negative, and PR negative, and Her2 negative
  Participants
    HR + | 21
    Triple Negative | 9
Prior lines of chemotherapy in the advanced setting [Median (Full Range); unit: line] | 1.5 [0 to 3]
PD-L1 positive cells [Count of Participants; unit: Participants]
  Positive | 4
  Negative | 21
  Missing sample | 4
  Specimen not adequate for evaluation | 1
TMB (mut/Mb) [Median (Full Range); unit: mut/Mb] — TMB: Tumor mutational burden
  mut/Mb | 10.9 [9 to 110]

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate of Nivolumab in Combination With Ipilimumab
Description: Overall Response Rate (ORR) is defined as the proportion of patients with complete or partial response evaluated by RECIST 1.1. Per RECIST 1.1: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Population: The analysis population includes all patients who initiated protocol therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 30
Participants | 5

2. Secondary Outcome: Overall Response Rate of the Combination According to Immune-related Response Criteria
Description: Overall Response Rate (ORR) is defined as the proportion of patients with complete or partial response evaluated by immune-related response criteria (irRC).
  Per irRC: irComplete Response (irCR): Complete disappearance of all tumor lesions (target an non-target) together with no new measurable/unmeasurable lesions for at least 4 weeks from the date of documentation of complete response.
  Immune-Related Partial Response (irPR): The sum of the products of the two largest perpendicular diameters of all target lesions is measured and captured as the SPD baseline. At each subsequent tumor assessment, the SPD of the two largest perpendicular diameters of all target lesions and of new measurable lesions are added together to provide the Immune Response Sum of Product Diameters (irSPD). A decrease, relative to baseline, of the irSPD compared to the previously SPD baseline of 50% or greater is considered an irPR.; Overall Response (OR) = irCR + irPR.
Time Frame: 2 years
Population: all patients who initiated protocol therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 30
Participants | 6

3. Secondary Outcome: Clinical Benefit Rate
Description: Clinical Benefit Rate (CBR) will be determined by looking at the number of subjects who have either a complete response, partial response, or stable disease for greater than or equal to 24 weeks, per RECIST 1.1
Time Frame: 2 Years
Population: analysis population includes all patients who initiated protocol therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 30
Participants | 5

4. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined from the study entry to first documented evidence of disease progression by RECIST 1.1 or death of any cause, whichever occurs first. Patients alive with no progression are censored at the last disease assessment.
Time Frame: 2 years
Population: all patients who initiated protocol therapy
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 30
month | 1.4 [1.3 to 4.6]

5. Secondary Outcome: Overall Survival
Description: OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Time Frame: Participants were followed long-term for survival every 12 weeks from the end of treatment until death or lost to follow-up. Median follow-up in this study cohort was 9.7 months.
Population: All patients who initiated protocol therapy
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 30
month | 19.3 [5.2 to NA] — Follow-up is not long enough/data is not mature to provide upper bound confidence interval.

ADVERSE EVENTS:
Time Frame: AE data were collected every cycle from the time of the first dose of the study treatment, through the end of the treatment. Vital status was followed even after patients were off treatment. AEs, including overall mortality, were observed up to 30 months.
Arm/Group | Nivolumab+Ipilimumab
All-Cause Mortality (participants affected / at risk) | 13/30
Serious Adverse Events (participants affected / at risk) | 5/30
Other Adverse Events (participants affected / at risk) | 24/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab+Ipilimumab (N=30)
Anorexia (Metabolism and nutrition disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac troponin T increased (Investigations) | 1
Confusion (Psychiatric disorders) | 1
Eyelid function disorder (Eye disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Lethargy (Nervous system disorders) | 1
Myasthenia gravis (Nervous system disorders) | 1
Myocarditis (Cardiac disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Platelet count decreased (Investigations) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab+Ipilimumab (N=30)
Anemia (Blood and lymphatic system disorders) | 3
Hypothyroidism (Endocrine disorders) | 2
Diarrhea (Gastrointestinal disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 2
Fatigue (General disorders and administration site conditions) | 9
Pain (General disorders and administration site conditions) | 3
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT03789110/Prot_SAP_000.pdf